CLINICAL TRIAL: NCT02965417
Title: An Open-label, Multicenter, Phase 2 Trial Investigating Sym004 in Patients With Metastatic Colorectal Cancer and Acquired Resistance to Anti-EGFR Monoclonal Antibodies and Documented Mutation of Extra Cellular Domain of EGFR (ECD-EGFR)
Brief Title: Sym004 in Metastatic Colorectal Cancer and ECD-EGFR Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Symphogen made a business decision to no longer perform the clinical study.
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-11; 2016-000621-39 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Resistance to anti-EGFR monoclonal antibodies; Mutation of ECD-EGFR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — futuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sym004 (Experimental): All patients will receive a loading dose of Sym004, followed by weekly (q1w) infusions
  Interventions: Drug: Sym004

INTERVENTIONS:
Drug: Sym004 — Sym004 is a 1:1 mixture of two monoclonal antibodies (mAbs) which bind to two non-overlapping epitopes of the Epidermal Growth Factor Receptor (EGFR).

SUMMARY:
This is a single arm, phase 2, open-label, multicenter trial in patients with metastatic colorectal cancer (mCRC) and acquired resistance to anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (mAbs) and documented mutation of extra cellular domain EGFR (ECD-EGFR).

ELIGIBILITY:
Inclusion and Exclusion criteria have been removed due to Symphogen's business decision to no longer perform the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Best overall response (OR) assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | 1 year

IPD SHARING:
Plan to Share IPD: Undecided